CLINICAL TRIAL: NCT00683488
Title: Integrated Treatment of Alcohol and/or Marijuana Abuse for HIV-Infected Youth - Phase I
Brief Title: Integrated Treatment of Marijuana Abuse for HIV+ Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATN 069
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: Substance Abuse; Adolescent community reinforcement approach; Adolescent Risk Behavior Assessment; Child and Adolescent Services Assessment; Cognitive behavioral therapy; Cognitive Therapy Rating Scale; Individual behavior therapy; Individual cognitive problem solving; Motivational enhancement therapy; HIV-Positive Youth With Substance Abuse; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Focus groups with adolescents with SA (Substance Abuse) will be conducted at each site (one group with 5 to 6 adolescents per site) to provide information on the areas of the intervention in need of adaptation in order to reflect the context of HIV infection.
  Interventions: Behavioral: Focus Group
- 2 (Experimental): The first intervention trial will enroll 9 participants (3 participants per site). Exit interviews of participants will assess acceptability, feasibility, and relevance of the intervention. Quantitative assessments pre and post intervention using audio computer-assisted self-interviewing (ACASI) will document immediate changes in substance use, sexual risk, and adherence to medical care. Additional qualitative feedback from interviews with mental health providers and study coordinators will address feasibility, acceptability, and relevance of the intervention and its methods.
  Interventions: Behavioral: First Intervention Trial
- 3 (Experimental): The revised intervention will be implemented with 20 participants (6 to 8 at each site). Exit interviews with subjects and feedback from mental health providers and study coordinators will provide the same qualitative information as in the first intervention trial. Quantitative data on participant outcomes such as substance use, sexual risk, and adherence to medical care will be collected pre, post and 3 month post intervention through ACASI.
  Interventions: Behavioral: Intervention Trial 2

INTERVENTIONS:
Behavioral: Focus Group — Focus group using and collecting feedback on the CBT/CM intervention.
  Arms: 1
Behavioral: First Intervention Trial — Intervention will comprise of approximately 15 weekly sessions.
  * Exit interviews at the end of each session will assess acceptability, feasibility, and relevance of the intervention.
  * Quantitative assessment (ACASI) pre and post intervention will document immediate changes in substance use, sexual risk, and adherence to medical care.
  * Qualitative feedback from interviews with mental health providers and study coordinators will address acceptability and feasibility.
  Arms: 2
Behavioral: Intervention Trial 2 — Evaluations/assessments will be similar to those involved for the first intervention trial. Study participants will return for a follow-up visit 3 months after the last intervention session to complete the ACASI.
  Arms: 3

SUMMARY:
This is an exploratory study that will adapt and test a combined cognitive behavioral treatment and contingency management intervention for alcohol and/or marijuana abuse for use in HIV-infected adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 16-24 years (inclusive) at the time of informed consent/assent as determined by medical record review or verbal verification from referring professional
* HIV-infected and aware of their status as documented by medical record review or verbal verification from referring professional
* Receives services at one of the three participating ATN clinic site or their community partners
* A score of 2 or greater on the CRAFFT indicating possible alcohol or marijuana use problem or abuse
* Alcohol and/or Marijuana Use or Abuse Disorder as indicated by the SSPQ-X
* Appropriate for an outpatient or intensive outpatient level of care in accordance with the American Academy of Child and Adolescent Psychiatry practice parameters as decided by site mental health provider in consultation with Drs. Brown and Esposito-Smythers
* English-speaking
* Ability and willingness to provide informed consent/assent for study participation
* Satisfactorily understands the nature of the study and the informed consent process as documented by the Consent Form Comprehension Assessment Questionnaire

Exclusion Criteria:

* Presence of serious psychiatric symptoms (e.g., active hallucinations, thought disorder)
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior)
* Intoxicated or under the influence of alcohol or other substances at the time of study entry

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2008-04; Primary Completion 2010-08 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To adapt a developmentally appropriate CBT/CM intervention for alcohol and/or marijuana abuse for HIV+ youth, relevant to the context of chronic medical care, emotion dysregulation due to frequent co-morbid psychiatric disorders and sexual risk behavior. | 2 years
To evaluate the acceptability, feasibility, and effectiveness of the CBT/CM intervention for alcohol and/or marijuana abuse, adherence to medical care, emotion regulation, and safer sexual behavior. | 2 years

SECONDARY OUTCOMES:
To revise the CBT/CM intervention based on information obtained in Phase 1 (this protocol), prepare for Phase 2 (to be supported by NIH), and disseminate the treatment manual to the ATN sites. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Larry K. Brown, M.D., Study Chair — Adolescent Trials Network
Locations (3):
- United States (3):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Mount Sinai Medical Center, New York, New York
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — https://www.atnonline.org